CLINICAL TRIAL: NCT03962439
Title: Impact of Challenging Engagement on Cognition in Older Adults: A Clinical Trial
Brief Title: Impact of Challenging Engagement on Cognition in Older Adults
Acronym: engAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis of cognitive data from the first 50 participants indicated that there was not a significant effect of the intervention on any key outcome measures and that a small increase in sample size was unlikely to improve this.
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Southern Methodist University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU 072018-048; 1R56AG058253-01 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Change
Keywords: Aging; Cognition; Alzheimer's Disease; Memory; Engagement; Digital Photography; Older Adults; Neural Function; Neuroimaging; Active Learning
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Demand Photography (Experimental): A structured, high-demand photography course targeting 210 hours of engagement over 16 weeks.
  Interventions: Behavioral: High-Demand Photography
- Moderate-Demand Photography (Active Comparator): A structured, moderate-demand photography course targeting 210 hours of engagement over 16 weeks.
  Interventions: Behavioral: Moderate-Demand Photography
- At-Home Engagement Group (Placebo Comparator): Participation, alone at home, in tasks that are relatively low in intellectual engagement.
  Interventions: Behavioral: At-Home Engagement

INTERVENTIONS:
Behavioral: High-Demand Photography — The high-demand photography group will receive 2.5 hours of instruction, twice a week, in a structured high-demand digital photography course plus 10 hours per week working on a special project at the research site without any formal instruction.
  Other Names: Productive Engagement Group (High)
  Arms: High-Demand Photography
Behavioral: Moderate-Demand Photography — The moderate-demand photography group will receive 2.5 hours of instruction, twice a week, in a structured moderate-demand digital photography course plus 10 hours per week working on a special project at the research site without any formal instruction.
  Other Names: Productive Engagement Group (Moderate)
  Arms: Moderate-Demand Photography
Behavioral: At-Home Engagement — The placebo control group will engage, alone at home, in tasks that are relatively low in intellectual engagement such as listening to music and radio or completing work-books that rely primarily on activation of knowledge.
  Other Names: Placebo Control
  Arms: At-Home Engagement Group

SUMMARY:
The study will enroll 90 participants in the "Impact of Challenging Engagement" study and assign them to one of three groups: high-demand photography, moderate-demand photography, and active placebo. These initial groups will allow us to collect data and address the feasibility of converting the project into a full trial. Participants will participate in one of three different engagement conditions for 15 hours per week, based on successful results from the initial Active Interventions for the Aging Mind (AIM) study - approved by University of Texas Southwestern (UTSW) Institutional Review Board (IRB) #072010-144. In the Impact of Challenging Engagement study, the lab will expand on the results of the AIM study to determine if high-demand activities result in any observable brain changes when compared to moderate demand or placebo activities. Behavioral and neural measures of cognitive change will be assessed, providing considerable insight into mechanisms of change. Participants will be characterized thoroughly in terms of behavioral tests of cognitive function, and a subset of subjects who meet neuroimaging criteria will undergo a functional magnetic resonance imaging (fMRI) procedure.

DETAILED DESCRIPTION:
All older adults experience some degree of cognitive compromise as they age and approximately 32 percent of adults aged 85 and older suffer from Alzheimer's disease (AD). The Alzheimer's Association estimates that delaying the onset of AD symptoms by only five years would reduce the rate of incidence by 50 percent! The present clinical trial builds on a wealth of observational work and more recent experimental research conducted in the PI's lab, which suggests that an important element of maintaining cognitive vitality for life is sustained engagement in mentally-challenging activities. In a U.S. sample of cognitively normal adults, investigators recently demonstrated that older adults who were randomly assigned to learn digital photography, quilting, or both, in fast-paced, demanding classes for 15 hours per week for three months, showed enhanced episodic memory function-both at the end of the engagement period and, importantly, one year later (Park et al., 2014). The observed memory improvements were in comparison to two active control conditions that were low in new learning: a social engagement group that had fun but did not engage in active learning, and a placebo condition where participants worked on low-effort cognitive tasks that relied on use of previous knowledge. The investigators also found similar facilitation effects when older adults were trained to use many different applications on an iPad. The lab most recently reported that older participants who participated in high-effort engagement conditions showed an increase in neural efficiency, exhibiting a change in neural activity from a pre-intervention pattern characteristic of older adults to a post-intervention pattern typical of young adults. Based on these findings, which included relatively small numbers of subjects, the investigators will conduct a larger clinical trial to determine whether mentally challenging activities facilitate memory in cognitively normal adults via changes of neural structure and function. The investigators propose to conduct a clinical trial study that will (a) evaluate the efficacy of different types of engagement in improving cognitive function in older adults, (b) examine the likelihood that mental effort invested is the underlying mechanism accounting for engagement effects, (c) show whether engaging in high-demand activities results in reliable brain changes. The investigators expect to demonstrate that when older adults engage for a sustained period of time in high-effort tasks (learning photography), both their memory and the modulation capacity of their brain will increase.

Randomization Procedure and Statistical Analyses:

Potential participants will complete an initial eligibility form. The investigators will contact those who are deemed eligible, will follow up with a TICS cognitive phone interview screening, and provide the link to an on-line demographic enrollment questionnaire.

The investigators will invite subjects who pass these screens to attend an informational session. At these sessions, project RAs will consent potential participants and have them complete the MRI screening form. The investigators will schedule consenting participants for cognitive testing and MRI scans (if applicable).

During the 3-week period set aside for cognitive and MRI testing, subjects will be assigned among the three treatment arms using a centrally created randomization scheme. Because baseline data for all potential participants will be available at the time of randomization, the rerandomization method of Morgan and Rubin (2012 Annals of Statistics 40:1263) will be utilized, which can achieve improved covariate balance in this setting. The investigators will generate a series of randomizations and evaluate them for balance on age, education, and sex, designating balance in terms of the MANOVA F statistic comparing the distributions of the covariates across the treatment groups. Once a randomization that meets this criterion is identified, it will be applied to the eligible participants.

Preliminary Analyses. In initial analyses, we will summarize categorical variables by proportions and continuous variables by means and quantiles. We will graph continuous variables and assess them for skewness, transforming if necessary (for example by logs or square roots) to render them more nearly normally distributed. We will explore relationships among variables by examining scatter plots and correlation matrices. We will conduct all analyses in R (version 3.3.2 or later) or SAS (version 9.4 or later).

Analysis of Primary Outcome Variables. The primary cognitive outcome endpoint will be a composite, scalar episodic memory score, as described in earlier research from the SYNAPSE project (5). This measure will exhibit substantial between-subject variability, in that subjects who give high scores at baseline are likely to give high scores at follow-up as well. To account for this, in primary analyses we will adjust for baseline levels by analysis of covariance - i.e., including baseline values together with treatment arm in a regression model for the post-treatment outcome. Alternatively (and equivalently), we can analyze the outcome variable in a mixed model, evaluating a treatment effect by estimating a time-by-treatment interaction. We will moreover conduct mixed-model analyses including the intermediate (6-week, mid-treatment) and long-term (1-year) values of the cognitive outcomes together with the end-of-treatment (12-week) outcome. As a secondary analysis to further elucidate the magnitude and timing of treatment effects, we will seek to create parsimonious models of this outcome as a function of time, treatment arm, stratification factors (center, age, sex, education) and potentially other factors measured at baseline. The primary brain outcome will be a vector measure of fMRI activation in four brain regions of interest, as described above and in previous work from SYNAPSE (7). This measure is also likely to exhibit substantial between-subject variability. We will again analyze the outcome variable in a mixed model, evaluating the treatment effect by estimating a time-by-treatment interaction, and conduct a secondary analysis where we model activation in the four regions as functions of time, treatment arm, stratification factors (center, age, sex, education) and potentially other factors measured at baseline.

Analysis of Secondary Outcomes. Dose-response. We anticipate that there will be a dose-response relationship, with the control arms having the lowest values, high-engagement arms, the highest values, and moderate-engagement arms having values in between. We will construct mixed models to estimate the sizes of these effects, and to determine whether effects are linear or nonlinear in the degree of engagement.

Subgroup Analyses. We will conduct a number of analyses aimed at estimating treatment effects within strata of age (younger or older than age 72), gender (male or female), education (greater or less than 14 years), and center (Dallas or Hamburg). We expect each of these strata to comprise roughly half of the subjects, except that our sample will likely be 65% female, reflecting the sex imbalance in the elderly. We will replicate our main analyses in each of the stratum subgroups, and additionally test for interactions.

Incomplete data. A major concern in any follow-up study is that there will be substantial dropout, eroding trial power. As indicated above, we expect no more than 15% to 20% of subjects to fail to complete the followup evaluation schedule. This is not a large fraction of dropout, and we have provided for its effects on power in our sample-size calculations. A second concern is that dropouts may differ systematically from completers, potentially introducing bias into estimated treatment contrasts. Our primary approach to analysis is to use mixed models, which give correct results as long as the dropout mechanism is missing at random - i.e., the probability of dropout, given the potentially missing observation and all prior observed data, does not depend on the potentially missing observation. Moreover, as long as the dropout is roughly balanced between treatment arms, it is unlikely to have a substantial biasing effect on estimated treatment effects, even if the dropout mechanism is not missing at random. In any event, if dropout is excessive or is unbalanced between arms, or there is concern that it is not missing at random, we are prepared to conduct analyses for sensitivity to nonignorable (i.e., biasing) dropout using general methods that Dr. Heitjan has developed.

Latent Factor Modeling. As a further form of secondary analysis, we will analyze the cognitive outcome variables simultaneously using a latent-variable approach. With this method, one models the several cognitive variables at each measurement time as being statistically independent given an unobserved, subject-specific latent variable. One accommodates serial correlation within subjects by estimating correlation of the latent variable within subjects over time. The approach evaluates treatment and time effects by modeling the mean of the latent variable as a function of the predictors, and each subject's estimated latent trajectory serves as a summary of his outcome status. We will also apply such models to the four-variate fMRI primary outcome.

Neuroimaging Analyses. We will test for a Group x Time interaction on the primary measure of modulation capacity. For the large-scale brain network analyses, we will utilize measures of connectivity between major nodes within the networks as indicators to develop constructs for the executive fronto-parietal network, salience network, and default network at each interval of data collection. To measure increases in hippocampal volume, we will segment the left and right hippocampus into four regions of interest (subiculum, CA1 and CA2/CA3/CA4, dentate gyrus, and entorhinal cortex) for all individual high-resolution MRI images. This division into 4 regions of interest (ROI) will ensure sufficient reliability and reproducibility of the subfield distinctions. These ROIs will be entered into the same Group x Time ANOVA as in the fMRI analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults at least 60 years old.
* At least 35 percent of participants will be men, and at least 15 percent will be minorities.
* 10th grade education or higher is required
* Fluent in English
* Alzheimer's Disease Assessment Scale-Cognitive (ADAS-COG) score of zero (a perfect score).
* A score of 18 or higher on the Barthel Index of Daily Functioning.
* Right-handed for magnetic resonance imaging (MRI) scanning.

Exclusion Criteria:

* Telephone Interview for Cognitive Status (TICS) lower than 25
* Montreal Cognitive Assessment (MOCA) score lower than 26
* Depression based on Center for Epidemiologic Studies Depression Scale (CESD) screening (a score of 27 or greater)
* Major psychiatric or neurological disorder
* Chemotherapy presently or in past year
* Coronary bypass presently or in past year
* History of major substance abuse
* History of central nervous system disease or brain injury
* Corrected vision poorer than 20/40 on Snellen Eye Chart after correction
* Recreational drug use in past six months
* Conditions which would contra-indicate MRI: Prior surgeries and/or implant of pacemakers, pacemaker wires, artificial heart valve, brain aneurysm surgery, middle ear implant, non-removable hearing aid or jewelry, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, artificial limb or joint; foreign metallic objects in the body such as bullets, ball-bullets or ball bearings (BB's), shrapnel, or metalwork fragments; pregnancy, vertigo, claustrophobia, left handedness, Body Mass Index (BMI) greater than 35, uncontrollable shaking, or inability to lie still for one hour.
* More than minimal experience with photography during the last 12 years
* Work at a structured job/volunteer more than 10 hours per week
* Computer experience that involves more than internet surfing and email
* Use of electronic devices to shop, pay bills, bank, and perform other higher-order functions
* Extensive experience with digital photography or post processing photo programs

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Park, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The engAGE Center: A Community Based Engagement Environment, Irving, Texas, United States

REFERENCES:
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Chan MY, Haber S, Drew LM, Park DC. Training Older Adults to Use Tablet Computers: Does It Enhance Cognitive Function? Gerontologist. 2016 Jun;56(3):475-84. doi: 10.1093/geront/gnu057. Epub 2014 Jun 13. PMID 24928557
- [Background] Park DC, Lodi-Smith J, Drew L, Haber S, Hebrank A, Bischof GN, Aamodt W. The impact of sustained engagement on cognitive function in older adults: the Synapse Project. Psychol Sci. 2014 Jan;25(1):103-12. doi: 10.1177/0956797613499592. Epub 2013 Nov 8. PMID 24214244
- [Background] Chan MY, Park DC, Savalia NK, Petersen SE, Wig GS. Decreased segregation of brain systems across the healthy adult lifespan. Proc Natl Acad Sci U S A. 2014 Nov 18;111(46):E4997-5006. doi: 10.1073/pnas.1415122111. Epub 2014 Nov 3. PMID 25368199

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Started | 17 | 15 | 18
Completed | 17 | 15 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data were analyzed from the first 50 participants, and then the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group | Total
Number analyzed (Participants) | 17 | 15 | 18 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 4 | 9
  >=65 years | 14 | 13 | 14 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.71 (4.07) | 68.20 (6.05) | 69.72 (5.19) | 68.92 (5.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 14 | 36
  Male | 6 | 4 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 7
  White | 15 | 13 | 13 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Episodic Memory [Mean (Standard Deviation); unit: scores on a scale] — Cognitive function will be measured using an episodic memory composite score. This score is composed of three tasks that measure episodic memory: National Institutes of Health (NIH) Picture Sequence Memory Test, Woodcock-Johnson Memory for names, and Rey Auditory Verbal Learning Test. A normalized distribution of the dependent variables from these measures will be created by applying a rank-ordered and standardized Blom transformation, and then averaging these scores, which may result in a sample mean of 0. Higher scores on this construct indicate better episodic memory (range: -1.4 to 1.3).
  scores on a scale | 0.13 (0.69) | -0.09 (0.77) | -0.04 (0.63) | 0 (0.68)
Speed of Processing [Mean (Standard Deviation); unit: scores on a scale] — Speed of processing is a construct that measures how rapidly individuals can process information. This construct is composed of three task that measure speed: the Digit Comparison Task, WAIS Digit Symbol Task, and the NIH Toolbox Pattern Comparison Task. These scores were averaged using a standardized Blom transformation, which may result in a sample mean of 0. Higher scores on the overall index at baseline, reported here, indicate greater speed (range: -1.8 to 1.9).
  scores on a scale | 0.17 (0.95) | 0.15 (0.49) | -0.28 (0.89) | 0 (0.83)
Reasoning [Mean (Standard Deviation); unit: scores on a scale] — Reasoning involves an individual's ability to recognize novel patterns and to effectively use these patterns to solve similar problems. This construct included the following reasoning tasks: Raven's Progressive Matrices and Education Test Services Letter Sets. These scores were averaged using standardized Blom transformation to form an index, which may result in a sample mean of 0. The baseline scores are reported here with higher scores indicating better reasoning (range: -2.0 to 1.8).
  scores on a scale | 0.12 (0.74) | -0.08 (0.89) | -0.05 (0.89) | 0 (0.83)
Working Memory [Mean (Standard Deviation); unit: scores on a scale] — Working memory measures the ability of individuals to simultaneously manipulate and store information. The construct was comprised of two tasks that measure working memory: The NIH Toolbox List Sorting Task and the Letter-Number Sequencing Task. These scores were averaged using a standardized Blom transformation to form an index, which may result in a sample mean of 0. A greater baseline score would indicate better working memory (range: -1.8 to 1.9).
  scores on a scale | 0.18 (0.93) | 0.01 (0.99) | -0.19 (0.78) | 0.00 (0.89)
Crystallized Intelligence [Mean (Standard Deviation); unit: scores on a scale] — Crystallized intelligence provides an estimation of the participant's world or vocabulary-based knowledge. This construct was comprised of three tasks: ETS Advanced Vocabulary task, the Shipley Vocabulary task, and The National Adult Reading Test (NART). These scores were averaged using standardized Blom transformation to form an index, which may result in a sample mean of 0. A greater baseline score would indicate better crystallized intelligence (range: -2.3 to 2.0).
  scores on a scale | 0.12 (0.61) | -0.09 (1.23) | -0.04 (0.84) | 0.00 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Episodic Memory Function
Description: Cognitive function will be measured using an episodic memory composite score. This score is composed of three tasks that measure episodic memory: National Institutes of Health (NIH) Picture Sequence Memory Test, Woodcock-Johnson Memory for names, and Rey Auditory Verbal Learning Test. A normalized distribution of the dependent variables from these measures will be created by applying a rank-ordered and standardized Blom transformation to pretest and posttest scores. The transformed standardized scores will then be averaged to create the episodic memory composite score. Cronbach's alpha will be calculated to test the internal reliability of the episodic memory construct. These measurements will be taken at baseline, and then following the intervention at week 16. A greater change score (week 16 - baseline), which is reported here, would indicate improved episodic memory (range: -1.2 to 1.2).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
scores on a scale
  Baseline score | 0.13 (0.69) | -0.09 (0.77) | -0.04 (0.63)
  Week 16 score | 0.24 (0.77) | 0.28 (0.67) | 0.13 (0.72)
  Change score (Week 16 - Baseline) | 0.12 (0.42) | 0.38 (0.42) | 0.17 (0.51)
Statistical Analysis 1: Comparison: High-Demand Photography vs Moderate-Demand Photography vs At-Home Engagement Group; Repeated measures ANCOVA testing whether change in episodic memory from baseline to 16 weeks interacted with condition (Time x Condition); Test type: Other — Null-hypothesis significance testing; p = .211, ANCOVA — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for baseline age, sex, and education; F-value = 1.61

2. Primary Outcome: Mean Change in Neural Modulation Capacity - Primary Brain Outcome Measure
Description: Brain activity drawn from four brain regions associated with effortful processing and memory-cingulate, precuneus, intraparietal sulcus, and inferior temporal gyrus-will be measured using fMRI. The primary fMRI task involves making living/nonliving judgments to presented words. Participants view a series of 128 nouns for 2500 ms each and judge whether each noun refers to a living or non-living item with a button press (yes or no). Half the words are living and half non-living. Moreover, half of the items within each category are easy to classify (e.g., LION or RADIO) or hard to classify (e.g., VIRUS or ZOMBIE), based on the categorical ambiguity of the item. This task measures modulation capacity between ambiguous and non-ambiguous words, where high modulation reflects greater neural efficiency and low modulation reflects poorer neural efficiency. These measurements will be taken at baseline, and then following the intervention (16 weeks later).
Time Frame: Baseline and 16 weeks
Population: As described in more detail in the Limitations and Caveats section for this project, this study was terminated early. Because of the time-intensive nature of processing imaging data, data for this measure were not processed and could not be reported.
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Speed of Processing
Description: Speed of processing is a construct that measures how rapidly individuals can process information. In the digit comparison task, participants have 45s to decide whether two strings of numbers are the same or different. The dependent variable (DV) is the number of items compared correctly summed across sections. In the WAIS Digit Symbol Task, participants are shown nine geometric symbols that are each assigned a digit from 1-9. Participants are then presented with randomized digits and asked to draw the corresponding symbol below each digit as quickly as possible for 90s. The DV is the number of items matched correctly in 90s. The NIH Toolbox Pattern Comparison task asks participants to discern whether two side-by-side pictures are the same or not. The DV is the number of items correct in a 90s period. These scores were standardized and averaged using a Blom transformation, and a greater change score (week 16 - baseline), reported here, would indicate improved speed (range: -.7 to 1).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
scores on a scale
  Baseline score | 0.17 (0.95) | 0.15 (0.49) | -0.28 (0.89)
  Week 16 score | 0.27 (0.83) | 0.14 (0.64) | -0.02 (0.84)
  Change score (Week 16 - Baseline) | 0.11 (0.31) | -0.01 (0.36) | 0.26 (0.40)
Statistical Analysis 1: Comparison: High-Demand Photography vs Moderate-Demand Photography vs At-Home Engagement Group; Repeated measures ANCOVA testing whether change in speed of processing from baseline to 16 weeks interacted with condition (Time x Condition); Test type: Other — Null hypothesis significance testing; p = .203, ANCOVA — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for baseline age, sex, and education; F-value = 1.66

4. Secondary Outcome: Working Memory
Description: Working memory measures the ability of individuals to simultaneously manipulate and store information. The construct was comprised of two tasks that measure working memory: The NIH Toolbox List Sorting Task and the Letter-Number Sequencing Task. These scores were standardized and averaged using Blom transformation to form an index. A greater change score (week 16 - baseline), reported here, would indicate improved working memory (range: -1.3 to 1).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
scores on a scale
  Baseline score | 0.18 (0.93) | 0.01 (0.99) | -0.19 (0.78)
  Week 16 score | 0.21 (0.85) | -0.17 (0.88) | -0.04 (1.02)
  Change score (Week 16 - baseline) | 0.03 (0.62) | -0.18 (0.41) | 0.15 (0.55)

5. Secondary Outcome: Reasoning
Description: Reasoning involves an individual's ability to recognize novel patterns and to effectively use these patterns to solve similar problems. In the Raven's Progressive Matrices task, participants are presented with visual patterns that have one piece missing and must determine which pattern out of 6 or 8 options is required to complete the visual pattern. Participants completed 24 problems, and the outcome is the number of items answered correctly in those 15 min. The ETS Letter Sets task involves presenting participants with 5 sets of letters, each set made up of 4 letters and being asked to determine which set of letters does not follow the same rule as the other 4 sets of letters. The outcome is number of items correct minus .25*(number of items incorrect). These scores were standardized and averaged using Blom transformation to form an index. A greater change score (week 16 - baseline), reported here, would indicate improved reasoning (range: -.7 to 1.5).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
scores on a scale
  Baseline score | 0.12 (0.74) | -0.08 (0.89) | -0.05 (0.89)
  Week 16 score | 0.31 (0.76) | 0.29 (0.84) | 0.19 (0.77)
  Change score (Week 16 - Baseline) | 0.18 (0.62) | 0.37 (0.35) | 0.24 (0.57)
Statistical Analysis 1: Comparison: High-Demand Photography vs Moderate-Demand Photography vs At-Home Engagement Group; Repeated measures ANCOVA testing whether change in reasoning from baseline to week 16 interacted with condition (Time x Condition); Test type: Other — Null hypothesis significance testing; p = .760, ANCOVA — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for baseline age, sex, and education; F-value = 0.28

6. Secondary Outcome: Crystallized Intelligence
Description: Crystallized intelligence provides an estimation of the participant's world or vocabulary-based knowledge. This construct was comprised of three tasks: ETS Advanced Vocabulary task, the Shipley Vocabulary task, and The National Adult Reading Test (NART). These scores were standardized and averaged using Blom transformation to form an index. A greater change score (week 16 - baseline), reported here, would indicate improved crystallized intelligence (range: -.7 to .7).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
scores on a scale
  Baseline score | 0.12 (0.61) | -0.09 (1.23) | -0.04 (0.84)
  Week 16 score | 0.13 (0.59) | 0.01 (1.12) | 0.07 (0.94)
  Change score (Week 16 - baseline) | 0.003 (0.37) | 0.10 (0.24) | 0.12 (0.28)

7. Secondary Outcome: Large-scale Brain Measures
Description: The procedures previously described in Chan et al., 2014 will be used to get a single measure of resting-state system segregation (both at baseline and following the intervention). This measure is calculated as the difference between the mean magnitudes of between-system correlations from the within-system correlations as a proportion of mean within-system correlation. Values greater than 0 reflect relatively lower between-system correlations in relation to within-system correlations (i.e., stronger segregation of systems), and values less than 0 reflect higher between-system correlations relative to within-system correlations (i.e., diminished segregation of systems).
Time Frame: Baseline and 16 weeks
Population: as for outcome 2
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Radial Diffusivity
Description: Radial diffusivity measures axonal/myelin damage by assessing water diffusion perpendicular to white matter fibres. Increased diffusivity (as measured in eigenvalues) indicate greater demyelination and therefore lower neural integrity.
Time Frame: Baseline and 16 weeks
Population: as for outcome 2
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Axial Diffusivity
Description: Axial diffusivity measures water diffusion that is parallel to white matter fibres. In contrast to radial diffusivity, a decrease in the axial diffusivity metric (in eigenvalues) is indicative of axonal damage.
Time Frame: Baseline and 16 weeks
Population: as for outcome 2
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Fractional Anisotropy
Description: Fractional anisotropy ranges from 0 to 1, and describes the degree of anisotropy (the property of substances to exhibit variations in physical properties along different axes) of a diffusion process. A value of 0 means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. A value of 1 means that diffusion occurs only along one axis and is fully restricted along all other directions. This measure reflects fibre density, axonal diameter, and myelination in white matter.
Time Frame: Baseline and 16 weeks
Population: as for outcome 2
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: NIH Picture Sequence Memory Test
Description: This measure involves showing pictured objects and activities that are thematically related to participants. The pictures are then minimized and moved to boundary of the screen throughout the trial in their fixed spatial order until all of the pictures in the sequence have been displayed. The pictures are then removed from their boundary locations and placed in a random assortment in the center of the screen. Participants are asked to move the pictures back into the sequence demonstrated as accurately as possible. The scores for this task consist of the number of adjacent pairs of pictures remembered correctly over 3 learning trials, with higher scores indicating better performance (range: 1 to 28). These variables factor into the episodic memory composite score (Outcome 1).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: total remembered pairs
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
total remembered pairs
  Baseline score | 12.65 (7.14) | 14.73 (4.57) | 10.50 (6.81)
  Week 16 score | 10.59 (7.1) | 15.73 (6.90) | 10.11 (7.13)
  Change score (Week 16 - baseline) | -2.06 (7.09) | 1.00 (5.94) | -0.39 (5.32)

12. Secondary Outcome: Woodcock-Johnson Memory for Names
Description: Participants are shown illustrations of space creatures while being told names for each creature. Participants are asked to recall the names of the space creatures by pointing to their corresponding illustration. Starting with 1 space creature, each trial adds 1 space creature to the list until the participant reaches a total of 12 learned creatures. This task is scored as a sum of the correct responses, with higher scores indicating better performance (range: 23 to 71), and is a variable in the episodic memory composite score.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: total correct responses
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
total correct responses
  Baseline score | 46.53 (9.91) | 47.60 (11.27) | 48.50 (13.74)
  Week 16 score | 54.76 (12.32) | 52.47 (10.21) | 53.72 (11.66)
  Change score (Week 16 - baseline) | 8.24 (8.08) | 4.87 (7.66) | 5.22 (9.01)

13. Secondary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: The RAVLT is a test of verbal learning and declarative memory. During the test, 15 nouns are read aloud for 5 consecutive trials. Each trial is followed by a free recall test (participant is asked to recall the words that were just read to them). The sum of correctly recalled words across 5 trials is called the total raw score. On completion of Trial 5, an interference list of 15 words (List B) is presented, followed by a free recall test of that list. After a 20-min delay, the examinee is again required to recall the words from list A - this is called the delay raw score. The raw scores for total items recalled, at list 1 and list 5, and the total for the delay trials are reported below with higher scores indicative of better performance (range: 0 to 15), and are incorporated into the episodic memory composite score.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: total items recalled
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
Number analyzed (Participants) | 17 | 15 | 18
total items recalled
  Baseline trial 1 score | 5.94 (1.75) | 5.53 (1.92) | 5.56 (1.42)
  Week 16 trial 1 score | 6.24 (2.08) | 5.87 (1.89) | 5.78 (1.80)
  Trial 1 change score (Week 16 - baseline) | 0.29 (2.17) | 0.33 (1.63) | 0.22 (2.21)
  Baseline trial 5 score | 12.53 (1.81) | 10.53 (2.75) | 11.67 (2.00)
  Week 16 trial 5 score | 12.71 (1.80) | 11.93 (1.79) | 11.89 (1.88)
  Trial 5 change score (Week 16 - baseline) | 0.18 (1.78) | 1.40 (2.97) | 0.22 (1.66)
  Baseline delayed score | 9.24 (3.63) | 7.60 (3.42) | 9.11 (2.03)
  Week 16 delayed score | 9.35 (3.30) | 9.53 (3.29) | 9.89 (2.45)
  delayed change score (Week 16 - baseline) | 0.12 (3.98) | 1.93 (2.89) | 0.78 (2.37)

ADVERSE EVENTS:
Time Frame: Participants could report AEs during testing (baseline and 16 weeks) or via email to the experimenter.
Description: This was a minimal risk study with no invasive procedures, so no AEs were expected.
Arm/Group | High-Demand Photography | Moderate-Demand Photography | At-Home Engagement Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15 | 0/18

LIMITATIONS AND CAVEATS:
As reported above, initial analyses of the effect of the photography training manipulation on episodic memory, speed of processing, and reasoning did not meet our a priori two-tailed p < .05 threshold for statistical significance (observed p-values > .2), and so the study was terminated. No additional statistical analyses were performed and because of the time-intensive nature of processing imaging data, data for outcome measures 2 and 7-10 were not processed and could not be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT03962439/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT03962439/ICF_001.pdf